CLINICAL TRIAL: NCT01241760
Title: A Randomized, Open-Label, Phase 3 Study of Telaprevir Administered Twice Daily or Every 8 Hours in Combination With Pegylated Interferon Alfa-2a and Ribavirin in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Virus Infection
Brief Title: VX-950-C211 - A Dosing Regimen Study (Twice Daily Versus Every 8 Hours) of Telaprevir in Treatment-naïve Participants With Genotype 1 Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013711; OPTIMIZE-HCV (Other: Janssen Infectious Diseases BVBA); VX-950-C211 (Other: Janssen Infectious Diseases BVBA); 2010-021628-84 (EudraCT Number)
Record Dates: First submitted 2010-10-28; First posted 2010-11-16 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Genotype 1 Chronic Hepatitis C; Treatment Naive
Keywords: Genotype 1 chronic hepatitis C; VX-950-C211; VX-950; IL28B; Telaprevir; Hepatitis C; BID; Q8h; SOC
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; telaprevir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 T(q8h) / PR (Experimental): Telaprevir (T) 750 mg (2 oral tablets) every 8 hours for 12 weeks, in combination with pegylated interferon (P) and ribavirin (R)
  Interventions: Drug: Ribavirin; Drug: Pegylated interferon alfa-2a; Drug: Telaprevir
- 002 T(b.i.d.) / PR (Experimental): Telaprevir (T) 1125 mg (3 oral tablets) twice a day (every 10-14 hours) for 12 weeks, in combination with pegylated interferon (P) and ribavirin (R)
  Interventions: Drug: Ribavirin; Drug: Telaprevir; Drug: Pegylated interferon alfa-2a

INTERVENTIONS:
Drug: Ribavirin — Ribavirin (RBV) 1000-1200 milligram (mg) per day (weight dependent) twice daily regimen oral tablets for 24 or 48 weeks depending on the patient's treatment response at week 4
Drug: Telaprevir — 1125 mg (3 oral tablets) twice a day (every 10-14 hours) for 12 weeks
  Arms: 002 T(b.i.d.) / PR
Drug: Pegylated interferon alfa-2a — 180 microgram (µg) per week, subcutaneous injection, for 24 or 48 weeks Pegylated interferon alfa-2a 180 microgram (µg) per week subcutaneous injection for 24 or 48 weeks depending on the patient's treatment response at week 4
Drug: Telaprevir — 750 mg (2 oral tablets) every 8 hours for 12 weeks
  Arms: 001 T(q8h) / PR

SUMMARY:
The purpose of this study is to evaluate the effectiveness of telaprevir administered twice daily versus every 8 hours in combination with Peg-IFN-alfa-2a and ribavirin in treatment-naïve participants with chronic HCV genotype 1 infection.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all persons know the study drug assignment) multicenter study to evaluate the effectiveness of telaprevir administered orally as 1125 milligram (mg) twice daily versus 750mg every 8 hours in combination with Peg-IFN-alfa-2a, administered via intramuscular injection once a week, and ribavirin, administered as an oral tablet twice a day, in treatment-naïve study participants with chronic hepatitis C virus (HCV) genotype 1 infection.

Telaprevir will be given orally (by mouth) from Day 1 through Week 12 as 3 tablets (1125mg) twice daily or 2 tablets (750mg) every 8 hours. Peg-IFN-alfa-2a will be administered once a week as an injection under the skin (180 microgram/week) from Day 1 through Week 24 or 48 (based on the patient's treatment response on week 4). Ribavirin is administered orally (by mouth) twice daily from Day 1 through Week 24 or 48 (based on the participant's treatment response on week 4) as 1,000-1,200 mg per day. After the end of treatment (Week 24, Week 48, or at early discontinuation of all study drugs), participants with undetectable HCV RNA at end of treatment will be required to attend follow-up visits until Week 72 safety/tolerability assessments will be performed throughout the treatment period and during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic HCV infection genotype 1 with HCV RNA level > 1,000 IU/mL
* Patients should not have had any previous treatment for hepatitis C
* Patient must have documentation of a liver biopsy within 2 years before the screening visit or the patient must agree to have a biopsy performed within the screening period
* Patients with cirrhosis should have serum alpha-fetoprotein (AFP) <= 50 ng/mL. If AFP > 50 ng/mL, absence of a mass must be demonstrated by ultrasound within the screening period
* A female patient of childbearing potential and a nonvasectomized male patient who has a female partner of childbearing potential must agree to the use of 2 effective methods of birth control from screening until 6 months (female patient) or 7 months (male patient) after the last dose of RBV.

Exclusion Criteria:

* Patient is infected or co-infected with HCV of another genotype than genotype 1 and/or patient is infected with more than one genotype subtype
* Patient has a pre-existing psychiatric condition
* Patient has history of decompensated liver disease or shows evidence of significant liver disease in addition to hepatitis C
* Patient has human immunodeficiency virus (HIV) or hepatitis B virus (HBV) co-infection
* Patient has active malignant disease or history of malignant disease within the past 5 years (with the exception of treated basal cell carcinoma).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (99):
- United States (37):
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Bradenton, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Downers Grove, Illinois
  - New Orleans, Louisiana
  - Lutherville, Maryland
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Egg Harbor Twp, New Jersey
  - Santa Fe, New Mexico
  - New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
- Australia (8):
  - Adelaide
  - Camperdown
  - Clayton
  - Darlinghurst
  - Fitzroy
  - Greenslopes
  - Melbourne
  - Perth
- Austria (3):
  - Graz
  - Linz
  - Vienna
- Belgium (6):
  - Antwerp
  - Brussels
  - Genk
  - Ghent
  - Leuven
  - Liège
- Brazil (4):
  - Campinas
  - Salvador
  - Santo André
  - São Paulo
- France (9):
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Lyon
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (8):
  - Berlin
  - Bochum
  - Essen
  - Frankfurt
  - Hamburg
  - Kiel
  - Mainz
  - Regensburg
- Dublin, Ireland
- Mexico (3):
  - Mex Ctity
  - México
  - Monterrey
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Kielce
  - Krakow
  - Warsaw
- Spain (6):
  - Barcelona
  - Madrid
  - Málaga
  - Santander
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Malmo
  - Stockholm
- United Kingdom (5):
  - Birmingham
  - Edinburgh
  - Glasgow
  - London
  - Manchester

REFERENCES:
- [Derived] Sarrazin C, Dierynck I, Cloherty G, Ghys A, Janssen K, Luo D, Witek J, Buti M, Picchio G, De Meyer S. An OPTIMIZE study retrospective analysis for management of telaprevir-treated hepatitis C virus (HCV)-infected patients by use of the Abbott RealTime HCV RNA assay. J Clin Microbiol. 2015 Apr;53(4):1264-9. doi: 10.1128/JCM.03030-14. Epub 2015 Feb 4. PMID 25653396
- [Derived] Buti M, Agarwal K, Horsmans Y, Sievert W, Janczewska E, Zeuzem S, Nyberg L, Brown RS Jr, Hezode C, Rizzetto M, Parana R, De Meyer S, De Masi R, Luo D, Bertelsen K, Witek J. Telaprevir twice daily is noninferior to telaprevir every 8 hours for patients with chronic hepatitis C. Gastroenterology. 2014 Mar;146(3):744-753.e3. doi: 10.1053/j.gastro.2013.11.047. Epub 2013 Dec 4. PMID 24316262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the effectiveness of telaprevir administered twice daily versus every 8 hours in combination with pegylated interferon and ribavirin in treatment-naïve participants with chronic HCV genotype 1 infection.
Pre-assignment Details: The study was conducted between 15 November 2010 and 02 August 2012 and recruited participants from 125 study centers in 14 countries worldwide. 744 participants were initially enrolled and 740 out of them randomly allocated to the 2 treatment arms.
Groups:
- T12(q8h)/PR: Telaprevir 750 mg (2 oral tablets) every 8 hours for 12 weeks, in combination with pegylated interferon (Peg-IFN)-alfa-2a solution for subcutaneous injection at the dose of 180 microgram per week (mcg/week) and ribavirin (RBV) oral tablets at the dose of 1000-1200 mg/day for 24 or 48 weeks depending on the treatment response at week 4.
- T12(b.i.d.)/PR: Telaprevir 1125 mg (3 oral tablets) twice a day (every 10-14 hours) for 12 weeks, in combination with pegylated interferon (Peg-IFN)-alfa-2a solution for subcutaneous injection at the dose of 180 microgram per week (mcg/week) and ribavirin (RBV) oral tablets at the dose of 1000-1200 mg/day for 24 or 48 weeks depending on the treatment response at week 4.
Period: Overall Study
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Started | 371 | 369
Completed | 337 | 329
Not Completed | 34 | 40
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 18 | 22
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Switch To Commercially Available Medicat | 1 | 4
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR | Total
Number analyzed (Participants) | 371 | 369 | 740
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 351 | 362 | 713
  >=65 years | 17 | 7 | 24
Age, Continuous [Mean (Full Range); unit: years] | 48 [18 to 70] | 47.5 [19 to 70] | 47.7 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 160 | 296
  Male | 235 | 209 | 444
Region of Enrollment [Number; unit: participants]
  Europe | 192 | 179 | 371
  North-America | 126 | 137 | 263
  Australia | 28 | 28 | 56
  Mexico | 5 | 4 | 9
  Brazil | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After the Last Planned Dose of Study Drugs (SVR12 Planned)
Description: The table below shows the percentage of participants achieving Sustained Virologic Response 12 weeks after last planned dose of study medication (SVR12 planned). SVR was defined as having Hepatitis C Virus (HCV) ribonucleic acid (RNA) levels less than 25 international units/milliliter (IU/mL).
Time Frame: End of trial, 12 weeks after last planned dose
Population: All analyses were performed on the full analysis (FA) set, which was defined as all randomized subjects who received at least one dose of study drug.
Measure: Number; unit: percentage of participants with response
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants with response | 72.8 | 74.3
Statistical Analysis 1: Comparison: T12(q8h)/PR vs T12(b.i.d.)/PR; Test type: Non-Inferiority or Equivalence — If the lower limit of the 95% confidence interval of the difference in proportions was above the pre-determined non-inferiority margin of -11%, non-inferiority was established; Regression, Logistic; The 95% confidence interval of the difference in proportions was estimated using a logistic regression model; Difference in proportion of response, % = 1.5, 95% CI [-4.9 to 12] — Observed data

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After the Last Planned Dose of Study Drugs (SVR24 Planned)
Description: The table below shows the percentage of participants achieving SVR 24 weeks after the last planned dose of study medication. SVR was defined as having Hepatitis C Virus (HCV) ribonucleic acid (RNA) levels less than 25 international units/milliliter (IU/mL). The response for T12(b.i.d)/PR group is higher than that after 12 weeks because HCV RNA data for two participants were missing for SVR assessment at that time. Consequently, by definition of SVR12, they were counted as not having achieved SVR12.
Time Frame: End of trial, 24 weeks after last planned dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants with response
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants with response | 72.8 | 74.8

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 72 Weeks After the Start of Study Medication (SVR72 Planned)
Description: The table below shows the percentage of participants achieving SVR 72 weeks after the start of study medication (SVR72 planned). SVR was defined as having plasma Hepatitis C Virus (HCV) ribonucleic acid (RNA) levels less than 25 IU/mL, target not detected, at end of treatment and up to 72 weeks after start of study medication (i.e., no confirmed detectable HCV RNA in between).
Time Frame: End of trial, 72 weeks after the start of study medication
Population: as for outcome 1
Measure: Number; unit: percentage of participants with response
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants with response | 69.0 | 70.2

4. Secondary Outcome: Percentage of Participants Achieving Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values of Less Than 25 IU/ml, Target Not Detected, at Different Time Points.
Description: The table below shows the percentage of participants with undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) levels, which means less than 25 IU/ml, target not detected, at different time points during the study.
Time Frame: Baseline, Week 4 and Week 4+12.
Population: as for outcome 1
Measure: Number; unit: percentage of participants with response
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants with response
  Baseline | 0 | 0
  at Week 4 | 67.4 | 69.4
  at Week 4 and Week 12 | 63.1 | 66.1

5. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure Which Required Them to Permanently Discontinue All Study Drugs
Description: The table below shows the percentage of participants who met a stopping rule, defined as having a hepatitis C virus (HCV) ribonucleic acid (RNA) value at Week 4 >1000 IU/mL and at Weeks 12, 24, 32 and 40 ≥25 IU/mL.
Time Frame: Week 4, 12, 24, 32, 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants | 9.7 | 10.3

6. Secondary Outcome: Percentage of Participants Who Relapsed During Follow-up Period
Description: The table below shows the percentage of participants who relapsed (ie, those having confirmed detectable hepatitis C virus [HCV] ribonucleic acid [RNA] during the 12-week follow-up period after previous HCV RNA <25 IU/mL, target not detected, at end of treatment).
Time Frame: During Follow-Up (24 weeks after the last dose of study drug)
Population: The analysis was performed on subjects with HCV RNA <25 IU/mL at the planned end of treatment, which included all randomized participants who received at least one dose of study drug and had data at the follow-up visit performed 24 weeks after the last dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 293 | 300
percentage of participants | 7.2 | 7.7

7. Secondary Outcome: Percentage of Participants of Each IL28B Genotype Achieving Sustained Virologic Response 12 Weeks After the Last Planned Dose of Study Medication (SVR12 Planned)
Description: The table below shows the effect of interleukin 28B (IL28B) gene's subtype (CC, CT or TT genotype) on the primary outcome measure: SVR12 planned.
Time Frame: End of trial, 12 weeks after the last planned dose
Population: as for outcome 1
Measure: Number; unit: percentage of participants with response
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR
Number analyzed (Participants) | 371 | 369
percentage of participants with response
  CC genotype (n = 108; n = 103) | 86.8 | 92.4
  CT genotype (n = 207; n = 207) | 67.8 | 67.5
  TT genotype (n = 56; n = 59) | 64.9 | 65.5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of study (12 weeks after the last dose).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Total: All
Arm/Group | T12(q8h)/PR | T12(b.i.d.)/PR | Total
Serious Adverse Events (participants affected / at risk) | 35/371 | 28/369 | 63/740
Other Adverse Events (participants affected / at risk) | 359/371 | 358/369 | 717/740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T12(q8h)/PR (N=371) | T12(b.i.d.)/PR (N=369) | Total (N=740)
Anaemia (Blood and lymphatic system disorders) | 14 | 13 | 27
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Abscess (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Asthenia (General disorders) | 1 | 1 | 2
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 3 | 2 | 5
Facial palsy (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Myoclonus (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Electrocardiogram t wave inversion (Investigations) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 1 | 2
Disorientation (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T12(q8h)/PR (N=371) | T12(b.i.d.)/PR (N=369) | Total (N=740)
Fatigue (General disorders) | 178 | 173 | 351
Pyrexia (General disorders) | 78 | 62 | 140
Asthenia (General disorders) | 72 | 65 | 137
Influenza like illness (General disorders) | 60 | 75 | 135
Chills (General disorders) | 43 | 22 | 65
Injection site reaction (General disorders) | 25 | 23 | 48
Pruritus (Skin and subcutaneous tissue disorders) | 158 | 158 | 316
Rash (Skin and subcutaneous tissue disorders) | 133 | 129 | 262
Dry skin (Skin and subcutaneous tissue disorders) | 35 | 43 | 78
Erythema (Skin and subcutaneous tissue disorders) | 22 | 20 | 42
Nausea (Gastrointestinal disorders) | 143 | 129 | 272
Diarrhoea (Gastrointestinal disorders) | 71 | 49 | 120
Anal pruritus (Gastrointestinal disorders) | 43 | 30 | 73
Vomiting (Gastrointestinal disorders) | 41 | 38 | 79
Anorectal discomfort (Gastrointestinal disorders) | 36 | 39 | 75
Haemorrhoids (Gastrointestinal disorders) | 33 | 26 | 59
Dry mouth (Gastrointestinal disorders) | 23 | 24 | 47
Dyspepsia (Gastrointestinal disorders) | 22 | 15 | 37
Proctalgia (Gastrointestinal disorders) | 21 | 18 | 39
Abdominal pain (Gastrointestinal disorders) | 19 | 10 | 29
Anaemia (Blood and lymphatic system disorders) | 148 | 155 | 303
Neutropenia (Blood and lymphatic system disorders) | 30 | 36 | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | 29 | 59
Headache (Nervous system disorders) | 108 | 87 | 195
Dysgeusia (Nervous system disorders) | 46 | 36 | 82
Dizziness (Nervous system disorders) | 30 | 41 | 71
Insomnia (Psychiatric disorders) | 68 | 69 | 137
Mood altered (Psychiatric disorders) | 47 | 37 | 84
Depression (Psychiatric disorders) | 36 | 27 | 63
Anxiety (Psychiatric disorders) | 20 | 26 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 39 | 83
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 36 | 71
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 41 | 33 | 74
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 25 | 49
Anorexia (Metabolism and nutrition disorders) | 36 | 30 | 66
Decreased appetite (Metabolism and nutrition disorders) | 19 | 22 | 41
Vision blurred (Eye disorders) | 17 | 20 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the PI (Investigator) wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.